CLINICAL TRIAL: NCT05495490
Title: Osseodensification Versus Osteotome Internal Sinus Lifting in Delayed Implant Placement (A Randomized Controlled Clinical Trial)
Brief Title: Osseodensification Versus Osteotome Internal Sinus Lifting in Delayed Implant Placement
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Omneya M. Elkadi, Assistant Lecturer, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FDASU-Rec ID032230; 1120 (Other: Ain Shams University)
Record Dates: First submitted 2022-08-05; First posted 2022-08-10 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Maxillary Sinus Floor Augmentation
Keywords: Osseodensification; Osteotome; Internal Sinus Lifting; Sticky Bone

STUDY DESIGN:
Intervention Model Description: Parallel single-blind masking randomized controlled clinical trial
Who Masked: Participant
Masking Description: Computer-generated randomization table
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Osseodensification Internal Sinus Lift / Sticky Bone graft material (Experimental): Osseodensification Internal Sinus Lift will be performed using sticky bone as a graft material.
  Interventions: Procedure: Osseodensification Internal Sinus Lift
- Osteotome Internal Sinus Lift /Sticky Bone graft material (Active Comparator): Osteotome Internal Sinus Lift will be performed using sticky bone as a graft material.
  Interventions: Procedure: Osteotome Internal Sinus Lift

INTERVENTIONS:
Procedure: Osseodensification Internal Sinus Lift — The osteotomy for the Osseodensification internal sinus lift begins with the advancement of a twist drill at 800 rpm and saline irrigation to within 1-2 mm of the sinus floor. The osteotomy is then widened by employing a series of osteotomy drills rotating at 800 rpm. Infracture of the sinus has occurred when the final osteotomy drill is advanced with gentle pressure at 100 rpm counterclockwise without irrigation until a bouncing sensation ("haptic feedback") occurs. After infracture, the graft material will be injected into the osteotomy site. Using the final osteotomy drill, the graft is guided apically. This procedure is repeated incrementally to raise the membrane. Once sufficient space has been created beneath the antral membrane, the implant will be inserted followed by suturing.
  Arms: Osseodensification Internal Sinus Lift / Sticky Bone graft material
Procedure: Osteotome Internal Sinus Lift — The osteotomy for the Osteotome internal sinus lift will begin with standard drills and saline irrigation to prepare the implant socket with a working length that is 1-2 mm shorter than the residual bone height as determined by radiographic examination. After preparation, a series of osteotomes of varying diameters will be sequentially utilized to widen the osteotomy and elevate the Schneiderian membrane by vertical tapping to create a "greenstick" fracture. The Valsalva maneuver (nasal blowing test) will be performed to determine the integrity of the Schneiderian membrane. During the osteotomy, the graft material will be injected and slowly placed into the elevated space using osteotomes until the desired depth is reached. Implant placement and suturing will conclude the procedure.
  Other Names: Bone-Added Osteotome Sinus Floor Elevation Technique; Summers Osteotome Technique
  Arms: Osteotome Internal Sinus Lift /Sticky Bone graft material

SUMMARY:
The sinus lift technique through alveolar crest Osseodensification is conservative, minimally invasive, and minimally traumatic, utilizing hydropneumatic counterclockwise rotating instruments to lift the maxillary sinus floor without touching the Schneiderian membrane, thereby minimizing the risk of perforation. In contrast, the internal sinus lift technique utilizing osteotomes to raise the Schneiderian membrane eliminated hammering, making the technique more patient-friendly, with the placement of a graft biomaterial around the implant. The challenge in this technique was the availability of > 5mm residual bone height preventing membrane perforation and low primary implant stability. Consequently, the investigator aims to compare the efficacy and clinical outcomes of Osseodensification and Osteotome internal sinus lifting after delayed implant placement by assessing bone gain and bone density around implants radiographically, the primary stability of the implants clinically, and patient satisfaction.

DETAILED DESCRIPTION:
Twenty patients with maxillary posterior edentulous ridge will be randomly assigned to one of two equal groups: Osseodensification sinus lift using sticky bone as a graft material (Group 1) and Osteotome internal sinus lift using sticky bone as a graft material (Group 2). (Group 2). Using Cone Beam Computed Tomography (CBCT), the sinus anatomy and height and width of the residual ridge from the sinus floor to the alveolar crest of all patients will be evaluated prior to surgery. Each patient will then receive pre-surgical medication consisting of intravenous steroidal anti-inflammatory drug (dexamethasone sodium phosphate 4mg) one hour prior to the procedure and oral rinsing with 0.12 percent chlorhexidine for one minute. After surgery, patients will receive 14 days of twice-daily chlorhexidine rinses 0.12 percent for postoperative treatment. Patients allergic to penicillin are given 1 g amoxicillin twice daily for six days or 0.5 g azithromycin. Ibuprofen (400) should be administered three times daily unless medically contraindicated. After insertion, the primary stability of each implant will be evaluated using a torque wrench and an Osstell device. All patients will undergo immediate postoperative CBCTs to assess bone gain and bone density. Utilizing the Visual Analogue Scale, patients' pain will be evaluated (VAS). A health-related quality of life questionnaire will be used to evaluate the patients' perception of recovery in terms of pain, oral function, general activity, and other symptoms. Postoperatively, the operator's subjective satisfaction with Osseodensification and Osteotome sinus lift techniques will be evaluated using a second printed questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patient partially edentulous with maxillary posterior edentulous ridge after extraction of more than 4 months.

  2. Both sexes will be selected males and females.

  3. Adult patients aged between 18 and 40 years of age.

  4. Good general health (American Society of Anesthesiology Physical Status Ⅰ-Ⅱ).

  5. Initial residual alveolar ridge height ranging between 4 to 6 mm according to preoperative CBCT.

  6. No previous surgery or radiation treatment on the maxillary sinus.

Exclusion Criteria:

* 1. Smokers.

  2. Pregnant or lactating females.

  3. Psychiatric disorders.

  4. Uncontrolled systemic disease.

  5. Hematologic diseases and coagulation disorders.

  6. Chemotherapy or radiotherapy of the head and neck area, and immunocompromised status.

  7. Medical conditions affecting bone metabolism and ongoing treatment with bisphosphonates drugs or systemic steroids.

  8. Presence of acute or chronic sinus pathoses or sinus membrane perforation.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-02-10 (Estimated); Primary Completion 2027-03-21 (Estimated); Study Completion 2027-04-21 (Estimated)

PRIMARY OUTCOMES:
Radiographic Assessment of Change in the Vertical Bone Height (Bone Gain). | Pre-operative and Immediately post-operative.
  The outcome will be obtained by the aid of Computed Cone Beam Tomography, assessing the amount of change from the pre-operative to the post-operative vertical bone height in millimeters.
Radiographic Assessment of Change in the Bone Density. | Pre-operative and Immediately post-operative.
  The outcome will be obtained by the aid of Computed Cone Beam Tomography assessing the amount of change from the pre-operative to the post-operative bone density values in Hounsfield unit.

SECONDARY OUTCOMES:
Clinical Assessment of Primary Stability of the Implants ( Insertion Torque Value) Measured by a Torque Wrench. | During procedure.
  The outcome will be obtained by the aid of a torque wrench and recorded in Newton centimeters.
  ( low torque (<30), medium torque (30 < Insertion Torque < 50), and high torque (>50).
Clinical Assessment of Primary Stability of the Implants (Implant Stability Quotient ) Measured by an Osstell® Device. | During procedure.
  The outcome will be obtained by the aid of an Osstell device, measured by the Resonance Frequency Analysis and determined by the Implant Stability Quotient ( within a 0-100 scale; 100 being maximum implant stability) .
Patient's Post-Operative Pain Assessment | 1 week post-operative
  The outcome will be obtained by the aid of a 100 mm Visual Analogue Scale (0 = minimal to; 100 = maximum)
Patient's Satisfaction Assessment. | 1 week post-operative
  The outcome will be obtained by the aid of a health-related quality of life questionnaire designed to assess the patient's perception of recovery concerning pain, oral function, general activity, and other symptoms.
Operator's Satisfaction Assessment | 1 year
  The outcome will be obtained by the aid of a a questionnaire assessing the operator's satisfaction with Osseodensification and Osteotome sinus lift techniques.

CONTACTS AND LOCATIONS:
Overall Officials: Hala A. Abuel- Ela, Professor, Study Director — Faculty of Dentistry- Ain Shams University; Mohamed W. Bissar, Lecturer, Study Director — Faculty of Dentistry- Ain Shams University; Omneya M. Elkadi, Principal Investigator — Faculty of Dentistry- Ain Shams University
Locations (2):
- Egypt (2):
  - Faculty of Dentistry- Assiut University, Asyut
  - Faculty of Dentistry- Ain Shams University, Cairo

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article after deidentification. (Text, tables, figures and appendices).
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Immediately following publication. No end date.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary identified for this purpose")

REFERENCES:
- [Background] Huwais S, Mazor Z, Ioannou AL, Gluckman H, Neiva R. A Multicenter Retrospective Clinical Study with Up-to-5-Year Follow-up Utilizing a Method that Enhances Bone Density and Allows for Transcrestal Sinus Augmentation Through Compaction Grafting. Int J Oral Maxillofac Implants. 2018 Nov/Dec;33(6):1305-1311. doi: 10.11607/jomi.6770. PMID 30427961
- [Background] Pjetursson BE, Lang NP. Sinus floor elevation utilizing the transalveolar approach. Periodontol 2000. 2014 Oct;66(1):59-71. doi: 10.1111/prd.12043. PMID 25123761
- [Background] Danesh-Sani SA, Loomer PM, Wallace SS. A comprehensive clinical review of maxillary sinus floor elevation: anatomy, techniques, biomaterials and complications. Br J Oral Maxillofac Surg. 2016 Sep;54(7):724-30. doi: 10.1016/j.bjoms.2016.05.008. Epub 2016 May 25. PMID 27235382
- [Background] Mourao CF, Valiense H, Melo ER, Mourao NB, Maia MD. Obtention of injectable platelets rich-fibrin (i-PRF) and its polymerization with bone graft: technical note. Rev Col Bras Cir. 2015 Nov-Dec;42(6):421-3. doi: 10.1590/0100-69912015006013. English, Portuguese. PMID 26814997
- [Background] Gheno E, Alves GG, Ghiretti R, Mello-Machado RC, Signore A, Lourenco ES, Leite PEC, Mourao CFAB, Sohn DS, Calasans-Maia MD. "Sticky Bone" Preparation Device: A Pilot Study on the Release of Cytokines and Growth Factors. Materials (Basel). 2022 Feb 16;15(4):1474. doi: 10.3390/ma15041474. PMID 35208017
- [Background] Zhou X, Hu XL, Li JH, Lin Y. Minimally Invasive Crestal Sinus Lift Technique and Simultaneous Implant Placement. Chin J Dent Res. 2017;20(4):211-218. doi: 10.3290/j.cjdr.a39220. PMID 29181458
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343